CLINICAL TRIAL: NCT05625880
Title: Evaluation of Bilirubin Estimates in Newborns From Smartphone Digital Images in a Nepali Population at Dhulikhel Hospital, Kathmandu University Hospital.
Brief Title: Evaluation of Bilirubin Estimates in Newborns From Smartphone Digital Images in a Nepali Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Picterus AS (Industry)
Collaborators: St. Olavs Hospital (Other); Dhulikhel Hospital (Other); National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Anders Aune, Chief medical officer, Picterus AS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2018/1608Nepal
Record Dates: First submitted 2022-11-10; First posted 2022-11-23 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Jaundice, Neonatal
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enable high qualitative estimation of bilirubin levels in the blood of new-borns (Experimental): There is only one arm in this study which is to enable high qualitative estimation of bilirubin levels in the blood of new-borns using Picterus JP.
  Interventions: Device: Picterus Jaundice Pro

INTERVENTIONS:
Device: Picterus Jaundice Pro — Use Picterus Jaundice Pro, a smartphone app that is used to take photo of the newborns skin, where the Picterus calibration card is place
  Other Names: Picterus JP

SUMMARY:
This cross-sectional study evaluates the accuracy of a novel smartphone application that estimates bilirubin levels in newborns at Dhulikhel Hospital, Kathmandu Nepal.

DETAILED DESCRIPTION:
This cross-sectional study evaluates the accuracy of a novel smartphone application that estimates bilirubin levels in 200 newborns at Dhulikhel Hospital, Kathmandu Nepal. The Picterus Calibration Card was placed on the chest of the newborn with the hole in the card placed over the infant's sternum. A validated smartphone with Picterus JP was used to collect digital images.

ELIGIBILITY:
Inclusion Criteria:

* Infants born with gestational age ≥35 weeks
* Birth weight ≥ 1750g
* Age 1 - ≤14 days
* Infants that will have a blood sample draw

Exclusion Criteria:

* Infants in the need for respiratory support
* Infants with conditions that could compromise skin circulation, as sepsis, heart failure
* Infants that have received phototherapy

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-08-06 (Actual)

PRIMARY OUTCOMES:
Enable high qualitative estimation of bilirubin levels in the blood of newborns, independent of skin color, using Picterus JP. | 5-10 minutes
  Evaluate of smartphone-based screening tool (Picterus JP) for neonatal jaundice in newborns at Dhulikhel Hospital, Kathmandu Nepal.

SECONDARY OUTCOMES:
correlation between bilirubin estimates in from a smartphone application and bilirubin measurements in serum in newborn | 1-2 hours
  To evaluate the correlation between bilirubin estimates in from a smartphone application and bilirubin measurements in serum in newborns with varying degree of jaundice
correlation between bilirubin estimates from a smartphone application and bilirubin estimates from a standard transcutaneous device in newborns | 5-10 minutes
  To evaluate the correlation between bilirubin estimates from a smartphone application and bilirubin estimates from a standard transcutaneous device in newborns with varying degree of jaundice
Correlation between bilirubin estimates from a smartphone application and bilirubin estimates from visual inspection in newborns | 5-10 minutes
  To evaluate the correlation between bilirubin estimates from a smartphone application and bilirubin estimates from visual inspection in newborns with varying degree of jaundice

CONTACTS AND LOCATIONS:
Overall Officials: Sunila Shakya, MD, PhD, Principal Investigator — Dhulikhel Hospital
Locations (1):
- Dhulikhel Hospital, Kathmandu University Hospital, Dhulikhel, Nepal